CLINICAL TRIAL: NCT01589978
Title: A U.S. Post-Approval Study of the PROMUS Element™ Plus Everolimus-Eluting Platinum Chromium Coronary Stent System
Brief Title: PROMUS Element Plus US Post-Approval Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2066
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stent; DES; atherosclerosis; everolimus
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Aspirin; Purinergic P2Y Receptor Antagonists; Clopidogrel; Ticlopidine; Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PROMUS Element (Experimental): Subjects who receive the PROMUS Element everolimus-eluting coronary stent
  Interventions: Device: PROMUS Element Plus Coronary Stent System; Drug: Aspirin; Drug: P2Y12 antagonist

INTERVENTIONS:
Device: PROMUS Element Plus Coronary Stent System — PROMUS Element is a device/drug combination product composed of two components, a device (coronary stent) and a drug product (a formulation of everolimus contained in a polymer coating).
  Other Names: PROMUS Element stent
Drug: Aspirin — Aspirin should be taken daily (81 mg) for 3 days prior to the procedure or as a peri-procedural loading dose of 250-500 mg. A maintenance dose of aspirin of at least 81 mg daily, or as indicated by the treating physician, should be continued indefinitely.
  Other Names: Acetyl salicylic acid
Drug: P2Y12 antagonist — Patients to take one of the following P2Y12 antagonists; maintenance doses to be continued per ACC/AHA/SCAI guidelines for PCI.
  * Clopidogrel: Per treating physician, peri-procedural loading dose (300-600 mg), subsequent maintenance dose (75 mg daily)
  * Prasugrel: Per treating physician, peri-procedural loading dose (60 mg), subsequent maintenance dose (10 or 5 mg daily per product labeling)
  * Ticagrelor: Per treating physician, peri-procedural loading dose (180 mg), subsequent maintenance dose (90 mg 2x daily); maintenance aspirin doses >100 mg may reduce ticagrelor effectiveness and should be avoided.
  * Ticlopidine: Per treating physician, if allergy/intolerance to clopidogrel, prasugrel, and/or ticagrelor, loading dose (500 mg), subsequent maintenance dose (250 mg 2x daily)
  Other Names: PLAVIX (clopidogrel); TICLID (ticlopidine); EFFIENT (prasugrel); BRILINTA (ticagrelor)

SUMMARY:
This study is designed to observe clinical outcomes in patients receiving the PROMUS Element Plus Everolimus-Eluting Platinum Chromium Coronary Stent System in routine clinical practice. Patients will have symptomatic heart disease or documented silent ischemia. This is a prospective, open-label consecutively-enrolling study. Clinical follow-up is through 5 years. Approximately 2,689 patients are to be enrolled in up to 65 centers in the United States.

DETAILED DESCRIPTION:
The wide-spread use of drug-eluting stents (DES) has evolved as standard of care in de novo lesions. The PROMUS Element Plus Everolimus-Eluting Platinum Chromium Coronary Stent System is indicated for improving luminal diameter in patients with symptomatic heart disease or documented silent ischemia due to de novo lesions in native coronary arteries ≥2.25 mm to ≤4.00 mm in diameter in lesions ≤34 mm in length. The proposed study will compile real-world clinical outcomes data for the PROMUS Element Plus Everolimus-Eluting Platinum Chromium Coronary Stent System in routine clinical practice.

Patients enrolled in this study are expected to follow antiplatelet therapy recommendations per American College of Cardiology (ACC)/American Heart Association (AHA)/Society for Cardiovascular Angiography and Interventions (SCAI) guidelines for percutaneous coronary intervention (PCI). Recommended medications include aspirin, which should be taken for 3 days prior to the procedure or as a peri-procedural loading dose and then continued indefinitely. Additionally, one of the following P2Y12 antagonists may be given in a peri-procedural loading dose and in a maintenance dose per physician discretion: clopidogrel, prasugrel, ticagrelor, or ticlopidine.

ELIGIBILITY:
Inclusion Criteria:

* The population will include consecutive, consented patients.

Exclusion Criteria:

* There are no exclusion criteria in this all-comers study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2681 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (52):
- United States (52):
  - Huntsville Hospital - The Heart Center, PC, Huntsville, Alabama
  - Springhill Medical Center, Mobile, Alabama
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Mercy General Hospital, Sacramento, California
  - Christiana Hospital, Newark, Delaware
  - Brandon Regional Hospital, Brandon, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Martin Memorial Health Systems - Martin Memorial Medical Center, Stuart, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Coliseum Medical Center, Macon, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Blessing Hospital, Quincy, Illinois
  - IU Health North Medical Center, Carmel, Indiana
  - Franciscan St. Francis Hospital, Indianapolis, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - St. Joseph Hospital, Lexington, Kentucky
  - Cardiovascular Research, LLC, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lakeland Hospitals at St. Joseph, Saint Joseph, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - North Memorial Medical Center, Minneapolis, Minnesota
  - United Hospital - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Forest County General Hospital, Hattiesburg, Mississippi
  - St. John's Regional Health Center (Springfield), Springfield, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Medical Center, New York, New York
  - St. Elizabeth Medical Center, Utica, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - St. Francis Hospital, Tulsa, Oklahoma
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University Medical Center-Greenville Memorial Hospital, Greenville, South Carolina
  - St. Francis Health System - St. Francis Hospital, Greenville, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - South Austin Hospital, Austin, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Chippenham Medical Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Meriter Hospital, Madison, Wisconsin
  - Marshfiled Clinic, Weston, Wisconsin

REFERENCES:
- [Derived] Beerkens FJ, Cao D, Batchelor W, Sartori S, Kandzari DE, Davis S, Tamis L, Wang JC, Othman I, Vogel B, Spirito A, Subramaniam V, Gigliotti OS, Haghighat A, Feng Y, Singh S, Lopez M, Giugliano G, Horwitz PA, Dangas G, Mehran R. Percutaneous Coronary Intervention in Men, Women, and Minorities With a Previous Coronary Artery Bypass Graft Surgery (from the Pooled PLATINUM Diversity and PROMUS Element Plus Registries). Am J Cardiol. 2023 Aug 1;200:204-211. doi: 10.1016/j.amjcard.2023.05.028. Epub 2023 Jun 22. PMID 37354778
- [Derived] Batchelor WB, Damluji AA, Yong C, Fiuzat M, Barnett SD, Kandzari DE, Sherwood MW, Epps KC, Tehrani BN, Allocco DJ, Meredith IT, Lindenfeld J, O'Connor CM, Mehran R. Does study subject diversity influence cardiology research site performance?: Insights from 2 U.S. National Coronary Stent Registries. Am Heart J. 2021 Jun;236:37-48. doi: 10.1016/j.ahj.2021.02.003. Epub 2021 Feb 24. PMID 33636137
- [Derived] Kandzari DE, Amjadi N, Caputo C, Rowe SK, Williams J, Tamboli HP, Christen T, Allocco DJ, Dawkins KD. One-Year Outcomes in "Real-World" Patients Treated With a Thin-Strut, Platinum-Chromium, Everolimus-Eluting Stent (from the PROMUS Element Plus US Post-Approval Study [PE-Plus PAS]). Am J Cardiol. 2016 Feb 15;117(4):539-545. doi: 10.1016/j.amjcard.2015.11.043. Epub 2015 Dec 7. PMID 26732420

RESULTS

PARTICIPANT FLOW:
Groups:
- PROMUS Element Overall Population: Subjects who receive the PROMUS Element everolimus-eluting coronary stent.
  Subgroups within the Overall Population Group:
  PLATINUM-Like Patients N=776 (at time of Primary endpoint)
  Defined as: all patients without acute MI, graft stenting, CTO, ISR, failed brachytherapy, bifurcation, ostial lesion, severe tortuosity, moderate or severe calcification by visual estimate in target lesion or target vessel proximal to target lesion, three-vessel stenting, cardiogenic shock, left main disease, or acute or chronic renal dysfunction (serum creatinine >2.0 mg/dl or patient on dialysis). For PLATINUM-like patients, lesion length and RVD should meet one of two criteria: 1) lesion length ≤28 mm and diameter ≥2.25 mm and <2.5 mm, or 2) lesion length ≤24 mm and diameter ≥2.5 mm and ≤4.25 mm.
  Long Lesion Patients N=340 Defined as: patients treated with at least one 32mm or 38mm (excluding patients only treated with 2.25 mm diameter and 32 mm length WH stent size) study stent.
Period: Overall Study
Arm/Group | PROMUS Element Overall Population
Started | 2681
Completed | 2681
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2681
Age, Continuous [Mean (Standard Deviation); unit: years] — Collected as part of a medical history during subject enrollment.
  years | 63.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Collected during subject enrollment.
  Participants
    Female | 807
    Male | 1874
Region of Enrollment [Number; unit: participants]
  United States | 2681
Cardiac History [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  Collected as part of a medical history during subject enrollment.
  participants
    History of CAD | 1625
    History of MI | 1409
    History of CHF | 275
    Stable Angina | 620
    Unstable Angina | 1347
    Silent Ischemia | 149
    History of PCI | 1159
    History of CABG | 457
Cardiac Risk Factors [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  Collected as part of a medical history during subject enrollment.
  participants
    Smoking, Ever | 1600
    Current Diabetic Mellitus | 989
    Hyperlipidemia Requiring Medication | 2016
    History of Hypertension Requiring Medication | 2077
    Family History of CAD | 1625
Lesion Characteristics: Target Lesion Vessel [Number; unit: lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Site reported information collected post-enrollment from medical records.
  lesions
    Left Anterior Descending Artery | 1339
    Circumflex Artery | 848
    Right Coronary Artery | 1165
    Left Main | 54
    Graft | 199
Lesion Characteristics: Lesion Length [Mean (Standard Deviation); unit: mm] — Site reported information collected post-enrollment from medical records.
  mm | 17.0 (10.3)
Lesion Characteristics: Reference Vessel Diameter [Mean (Standard Deviation); unit: mm] — Site reported information collected post-enrollment from medical records.
  mm | 2.94 (0.51)
Lesion Characteristics: Pre-Procedure Thrombolysis in Myocardial Invarction (TIMI) Flow [Number; unit: lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Site reported information collected post-enrollment from medical records. Stages range from TIMI 0 (no perfusion) to TIMI 3 (normal flow).
  TIMI: Thrombolysis in Myocardial Infarction
  lesions
    0 | 359
    1 | 157
    2 | 487
    3 | 2539

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death or Myocardial Infarction Rate in PLATINUM-like Patients
Description: Cardiac death or myocardial infarction rate at 12 months post implantation in PLATINUM-like patients (no acute myocardial infarction, graft stenting, chronic total occlusion, in-stent restenosis, failed brachytherapy, bifurcation, ostial lesion, severe tortuosity, moderate/severe calcification, 3-vessel stenting, cardiogenic shock, left main disease, or acute/chronic renal dysfunction; lesion length ≤28 mm with reference vessel diameter ≥2.25 mm and <2.5 mm, or lesion length ≤24 mm with diameter ≥2.5 mm and ≤4.25 mm); statistical testing will assess if rate meets the performance goal (3.2%)
Time Frame: 12 months
Population: Note: PLATINUM-like population for the Primary Endpoint at 12 months includes PROMUS Element patients from the PLATINUM trials (WH and SV) (N=862), PLATINUM-like patients from PE-Prove (N=269), and PLATINUM-like patients from PROMUS Element Plus US Post-Approval Study (N=776) (as stated as a subgroup in the Participant Flow Module.
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 1907
percentage of patients | 1.78
Statistical Analysis 1: Comparison: PROMUS Element; One-sided, single binomial test will be performed to compare observed rate against performance goal, the normal approximation of the test statistic will be used. The performance goal is met if the one-sided upper 95% confidence bound for the observed binary rate is less than performance goal; Test type: Non-Inferiority or Equivalence — Given the performance goal of 3.2%, with expected rate for PROMUS Element Plus of 2.2% and a one-sided 5% significance level, approximately 1,706 PLATINUM-like patients will provide at least 80% power to reject the null hypothesis if it is false; p < .0001, Chi-squared

2. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition in PLATINUM-like Patients
Description: ARC definite/probable ST rate in PLATINUM-like patients (no acute myocardial infarction, graft stenting, chronic total occlusion, in-stent restenosis, failed brachytherapy, bifurcation, ostial lesion, severe tortuosity, moderate/severe calcification, 3-vessel stenting, cardiogenic shock, left main disease, or acute/chronic renal dysfunction; lesion length ≤28 mm with reference vessel diameter ≥2.25 mm and <2.5 mm, or lesion length ≤24 mm with diameter ≥2.5 mm and ≤4.25 mm); statistical testing will assess if the annual ST rate increase after the first year meets the performance goal (1.0%)
Time Frame: 12 months
Population: PROMUS Element PLATINUM-Like patients (a subgroup of the overall population as described in the Participant Flow Module), N=776.
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 776
percentage of patients | 0.3

3. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition in All Patients
Description: DEFINITE ST: acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE ST: unexplained death within 30 days or target-vessel infarction without angiographic information ARC ST is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute ST: 0-24 hours after stent implantation; Subacute ST: >24 hours to 30 days post; late ST: >30 days to 1 year post; Very late ST: >1 year post; NOTE: Acute/subacute can be replaced by early ST (0-30 days)
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2681
percentage of patients | 0.7

4. Secondary Outcome: Rate of Longitudinal Stent Deformation
Description: Compression/elongation of a stent along its long axis resulting from interaction with an ancillary device (e.g., guide catheter) which catches the stent end or an internal stent strut; can occur with advancement or withdrawal of ancillary device. Under fluoroscopy, longitudinal compression usually results in increased strut density and elongation in decreased strut density ('pseudo-fracture'); both can occur in the same stent.
Time Frame: Index Procedure
Measure: Number; unit: stents
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2681
stents | 2

5. Secondary Outcome: Major Adverse Cardiac Event Rate (MACE)
Description: Composite of cardiac death, myocardial infarction, and target vessel revascularization
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 6.9

6. Secondary Outcome: Rate of Major Adverse Cardiac Events Related to the PROMUS Element Stent
Description: Composite of cardiac death, myocardial infarction, and target vessel revascularization related to the PROMUS Element stent
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 4.7

7. Secondary Outcome: Myocardial Infarction (MI) Rate
Description: New Q-waves in ≥2 leads lasting ≥0.04 sec with creatine kinase myoglobin band(CK-MB) or troponin >upper limit of normal(ULN); if no new Q-waves total CK levels >3×ULN (peri-percutaneous coronary intervention [PCI]) or >2×ULN (spontaneous) with elevated CK-MB or troponin >3×ULN (peri-PCI) or >2×ULN (spontaneous) plus ≥one of the following: ECG changes indicating new ischemia (new ST-T changes, left bundle branch block), imaging evidence of new loss of viable myocardium, new regional wall motion abnormality. Similar for MI diagnosis post coronary artery bypass graft with CK-MB or troponin >5×ULN
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 1.1

8. Secondary Outcome: Rate of Myocardial Infarction (MI) Events Related to the PROMUS Element Stent
Description: as for outcome 7
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 0.7

9. Secondary Outcome: Cardiac Death Rate
Description: Cardiac death is defined as death due to any of the following: acute myocardial infarction; cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident through hospital discharge or cerebrovascular accident suspected of being related to the procedure; death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery; any death in which a cardiac cause cannot be excluded
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 1.4

10. Secondary Outcome: Rate of Cardiac Death Events Related to the PROMUS Element Stent
Description: as for outcome 9
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 1.3

11. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Description: Target vessel revascularization is defined as any attempted or successfully completed percutaneous or surgical revascularization of a target vessel.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 5.6

12. Secondary Outcome: Rate of Target Vessel Revascularization (TVR) Events Related to the PROMUS Element Stent
Description: as for outcome 11
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 3.5

13. Secondary Outcome: Cardiac Death or Myocardial Infarction (MI) Rate
Description: See individual descriptions of events.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 2.3

14. Secondary Outcome: Rate of Cardiac Death or Myocardial Infarction Events Related to the PROMUS Element Stent
Description: See individual descriptions of events.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 1.8

15. Secondary Outcome: Target Vessel Failure (TVF) Rate
Description: Target vessel failure (TVF) is defined as any revascularization of the target vessel, myocardial infarction (MI) related to the target vessel, or death related to the target vessel.
  For the purposes of this protocol, if it cannot be determined with certainty whether MI or death was related to the target vessel it will be considered TVF.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 6.7

16. Secondary Outcome: Rate of Target Vessel Failure (TVF) Related to the PROMUS Element Stent
Description: as for outcome 15
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 4.7

17. Secondary Outcome: All Death Rate
Description: All death includes cardiac death and non-cardiac death.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 2.3

18. Secondary Outcome: Non-cardiac Death Rate
Description: Non-cardiac death is defined as death not due to cardiac causes.
  Cardiac death is death due to any of the following: acute myocardial infarction; cardiac perforation/pericardial tamponade; arrhythmia or conduction abnormality; cerebrovascular accident through hospital discharge or cerebrovascular accident suspected of being related to the procedure; death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery; any death in which a cardiac cause cannot be excluded.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 0.9

19. Secondary Outcome: All Death or Myocardial Infarction Rate
Description: See description of individual events.
Time Frame: ≤24 hours, 30 days, 180 days, annually through 5 years
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 2554
percentage of patients | 3.2

20. Secondary Outcome: Target Vessel Failure (TVF) Rate in PLATINUM-like Medically Treated Diabetic Patients
Description: Any revascularization of the target vessel, myocardial infarction related to the target vessel, or death related to the target vessel. See individual components for descriptions. Statistical testing will determine if the rate meets the performance goal (12.6%)
Time Frame: 12 Months
Measure: Number; unit: percentage of patients
Arm/Group | PROMUS Element
Number analyzed (Participants) | 276
percentage of patients | 3.26

21. Secondary Outcome: ARC ST Rate in PLATINUM-like Population.
Description: Using the Academic Research Consortium (ARC) definition, the (definite/probable) stent thrombosis (ST) rate in the PLATINUM-like* population will be analyzed. Statistical testing will be used to determine if the annual increase after the first year in ST rates observed in PLATINUM-like patients meets the performance goal of 1.0% (expected rate of 0.4% + a delta of 0.6%).
Time Frame: Annually through 5 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- PROMUS Element Overall Population: Subjects who receive the PROMUS Element everolimus-eluting coronary stent.
Arm/Group | PROMUS Element Overall Population
Number analyzed (Participants) | 1907
percentage of participants | 0.0023
Statistical Analysis 1: Comparison: PROMUS Element Overall Population; The expected annual increase of stent thrombosis rate is assumed to be 0.4%, based on the observed increase in incidence rate of stent thrombosis of approximately 0.4% annually for PLATINUM-like patients in the pooled TAXUS SR Express and pooled TAXUS Liberté data. Using a delta of 0.6%, the performance goal is set to 1.0% (expected rate + delta = 0.4% + 0.6% = 1.0%); Test type: Non-Inferiority or Equivalence — The sample size is calculated for one-sample chi-square test for a single proportion using nQuery AdvisorVersion 5.0. The expected annual increase in ST rate is estimated to be 0.4% based on the current data available from the pooled TAXUS Express and pooled TAXUS Liberté data and the PG is 1.0% using a delta of 0.6%. Given a one-sided 5% significance level, a minimum of 1,660 PLATINUM-like patients at 5-yrs will be required to provide 90% power to reject the null hypothesis if it is false; p < .0001, Chi-squared

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from the point of subject enrollment through primary endpoint (12 months).
Arm/Group | PROMUS Element
Serious Adverse Events (participants affected / at risk) | 780/2681
Other Adverse Events (participants affected / at risk) | 5/2681
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PROMUS Element (N=2681)
ANGINA PECTORIS (Cardiac disorders) | 120
ANGINA UNSTABLE (Cardiac disorders) | 93
CORONARY ARTERY DISEASE (Cardiac disorders) | 49
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 46
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 33
MYOCARDIAL INFARCTION (Cardiac disorders) | 22
ATRIAL FIBRILLATION (Cardiac disorders) | 23
CORONARY ARTERY DISSECTION (Cardiac disorders) | 19
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 15
ACUTE CORONARY SYNDROME (Cardiac disorders) | 10
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 10
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 8
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 7
CORONARY ARTERY STENOSIS (Cardiac disorders) | 7
CARDIOMYOPATHY (Cardiac disorders) | 6
CARDIAC ARREST (Cardiac disorders) | 5
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 5
CARDIOGENIC SHOCK (Cardiac disorders) | 4
ATRIAL FLUTTER (Cardiac disorders) | 3
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 3
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3
VENTRICULAR FIBRILLATION (Cardiac disorders) | 3
CARDIAC FAILURE (Cardiac disorders) | 2
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 2
POSTINFARCTION ANGINA (Cardiac disorders) | 2
SINUS BRADYCARDIA (Cardiac disorders) | 2
TACHYCARDIA (Cardiac disorders) | 2
AORTIC VALVE STENOSIS (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 1
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1
PALPITATIONS (Cardiac disorders) | 1
SICK SINUS SYNDROME (Cardiac disorders) | 1
SINUS ARRHYTHMIA (Cardiac disorders) | 1
TACHYARRHYTHMIA (Cardiac disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 78
DEATH (General disorders) | 9
CHEST PAIN (General disorders) | 8
ASTHENIA (General disorders) | 4
CHEST DISCOMFORT (General disorders) | 4
INFLUENZA LIKE ILLNESS (General disorders) | 2
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2
ULCER HAEMORRHAGE (General disorders) | 2
ADVERSE EVENT (General disorders) | 1
BLOODY DISCHARGE (General disorders) | 1
CATHETER SITE HAEMATOMA (General disorders) | 1
HERNIA (General disorders) | 1
IMPAIRED HEALING (General disorders) | 1
MALAISE (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
PAIN (General disorders) | 1
PYREXIA (General disorders) | 1
PNEUMONIA (Infections and infestations) | 36
CELLULITIS (Infections and infestations) | 9
SEPSIS (Infections and infestations) | 8
URINARY TRACT INFECTION (Infections and infestations) | 8
OSTEOMYELITIS (Infections and infestations) | 6
BRONCHITIS (Infections and infestations) | 5
UROSEPSIS (Infections and infestations) | 4
APPENDICITIS (Infections and infestations) | 3
BACTERAEMIA (Infections and infestations) | 3
DIVERTICULITIS (Infections and infestations) | 3
INFLUENZA (Infections and infestations) | 3
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 3
ABSCESS LIMB (Infections and infestations) | 2
BRONCHIECTASIS (Infections and infestations) | 2
GANGRENE (Infections and infestations) | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 2
INFECTION (Infections and infestations) | 2
LOBAR PNEUMONIA (Infections and infestations) | 2
WOUND INFECTION (Infections and infestations) | 2
ABDOMINAL ABSCESS (Infections and infestations) | 1
ANOGENITAL WARTS (Infections and infestations) | 1
BRONCHITIS VIRAL (Infections and infestations) | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
MYCOBACTERIAL INFECTION (Infections and infestations) | 1
OSTEOMYELITIS ACUTE (Infections and infestations) | 1
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 1
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1
PURULENT DISCHARGE (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 24
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 19
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 13
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 7
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 6
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 4
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 4
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
ALLERGIC BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
MEDIASTINAL MASS (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 15
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 5
DYSPHAGIA (Gastrointestinal disorders) | 5
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 5
COLITIS (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 4
GASTRIC ULCER (Gastrointestinal disorders) | 4
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3
MELAENA (Gastrointestinal disorders) | 3
PANCREATITIS (Gastrointestinal disorders) | 3
ABDOMINAL HERNIA (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Respiratory, thoracic and mediastinal disorders) | 2
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 2
GASTRITIS (Gastrointestinal disorders) | 2
GASTRITIS EROSIVE (Gastrointestinal disorders) | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 2
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 2
ANAL FISTULA (Gastrointestinal disorders) | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1
GASTRIC DISORDER (Gastrointestinal disorders) | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTRIC POLYPS (Gastrointestinal disorders) | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
INTESTINAL POLYP (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 1
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
SYNCOPE (Nervous system disorders) | 17
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 13
CAROTID ARTERY STENOSIS (Nervous system disorders) | 11
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 7
ENCEPHALOPATHY (Nervous system disorders) | 4
PRESYNCOPE (Nervous system disorders) | 3
CEREBRAL INFARCTION (Nervous system disorders) | 2
DYSARTHRIA (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 2
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2
BASAL GANGLIA INFARCTION (Nervous system disorders) | 1
BRAIN STEM STROKE (Nervous system disorders) | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1
CONVULSION (Nervous system disorders) | 1
ENCEPHALITIS (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
LETHARGY (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
RADICULAR PAIN (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 9
DEEP VEIN THROMBOSIS (Vascular disorders) | 8
HYPERTENSION (Vascular disorders) | 7
HYPOTENSION (Vascular disorders) | 7
AORTIC STENOSIS (Vascular disorders) | 4
ARTERIOSCLEROSIS (Vascular disorders) | 3
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 3
HAEMATOMA (Vascular disorders) | 3
PERIPHERAL ISCHAEMIA (Vascular disorders) | 3
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 3
HYPERTENSIVE CRISIS (Vascular disorders) | 2
MALIGNANT HYPERTENSION (Vascular disorders) | 2
ACCELERATED HYPERTENSION (Vascular disorders) | 1
AORTIC ANEURYSM (Vascular disorders) | 1
ARTERIAL THROMBOSIS (Vascular disorders) | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
ISCHAEMIA (Vascular disorders) | 1
ISCHAEMIC LIMB PAIN (Vascular disorders) | 1
LYMPHOEDEMA (Vascular disorders) | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1
PERIPHERAL COLDNESS (Vascular disorders) | 1
SHOCK (Vascular disorders) | 1
TAKAYASU'S ARTERITIS (Vascular disorders) | 1
THROMBOPHLEBITIS (Vascular disorders) | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 5
HIP FRACTURE (Injury, poisoning and procedural complications) | 4
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 2
DRUG TOXICITY (Injury, poisoning and procedural complications) | 2
FALL (Injury, poisoning and procedural complications) | 2
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 2
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 2
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 2
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2
RIB FRACTURE (Injury, poisoning and procedural complications) | 2
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1
ANASTOMOTIC ULCER HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1
DISLOCATION OF JOINT PROSTHESIS (Injury, poisoning and procedural complications) | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
SEROMA (Injury, poisoning and procedural complications) | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 1
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 1
WOUND (Injury, poisoning and procedural complications) | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 13
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 4
NEPHROLITHIASIS (Renal and urinary disorders) | 3
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 3
RENAL FAILURE (Renal and urinary disorders) | 3
URINARY RETENTION (Renal and urinary disorders) | 3
HAEMATURIA (Renal and urinary disorders) | 2
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 2
BLADDER OBSTRUCTION (Renal and urinary disorders) | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 1
RENAL DISORDER (Renal and urinary disorders) | 1
URETHRAL MEATUS STENOSIS (Renal and urinary disorders) | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ANAEMIA (Blood and lymphatic system disorders) | 11
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 6
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 1
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
DIABETIC FOOT (Metabolism and nutrition disorders) | 1
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
OBESITY (Metabolism and nutrition disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 4
CHOLECYSTITIS (Hepatobiliary disorders) | 3
GALLBLADDER DISORDER (Hepatobiliary disorders) | 2
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1
CHOLANGITIS (Hepatobiliary disorders) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1
BLOOD CREATININE INCREASED (Investigations) | 1
BLOOD GLUCOSE DECREASED (Investigations) | 1
BLOOD URINE (Investigations) | 1
CATHETERISATION CARDIAC (Investigations) | 1
ANXIETY (Psychiatric disorders) | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1
CONVERSION DISORDER (Psychiatric disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 3
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
DIVERTICULITIS MECKEL'S (Congenital, familial and genetic disorders) | 1
CATARACT (Eye disorders) | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1
CAROTID ENDARTERECTOMY (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PROMUS Element (N=2681)
Myocardial Infarction (Cardiac disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less